CLINICAL TRIAL: NCT01022814
Title: Development of a Diagnostic Device for Identifying Between Amniotic Fluid to Urine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Arik Tzukert, Hadassah Medical Organization
Other Study IDs: Momteclife-HMO-CTIL
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Color Reaction With Amniotic Fluid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Pregnant woman
  Interventions: Device: A disposable pad containing sensitive chemical indicators

INTERVENTIONS:
Device: A disposable pad containing sensitive chemical indicators — After a urine/amniotic fluid leaking, liquid meets the diagnostic device and chemical reactions will occur in the test zones and cause a color change.

SUMMARY:
In the final months of pregnancy, women need to know whether their 'water is broken' necessitating a race to the delivery room, or whether pressure of the foetus on their bladder has caused them merely to pass urine. They may also have faced the same dilemma on many occasions much earlier in the pregnancy. With this development the investigators will provide them with an immediate answer to this critical question.

ELIGIBILITY:
Inclusion Criteria:

* Amniotic fluid that were taken after the 17th week.

Exclusion Criteria:

* None.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: An unrecognized amniotic fluid that passed a genetic analysis and appointed to be disposed.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nili Yanai, Dr', Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel